CLINICAL TRIAL: NCT01961388
Title: Study to Assess the Dietary Carbohydrate Content of Indian Diabetics With Special Therapeutic View on Effectiveness of Acarbose and Metformin Monotherapy
Acronym: STARCH AM
Status: Withdrawn | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16667; GB1311IN (Other: company internal)
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Acarbose_BAY G5421
  Interventions: Drug: Bay G5421 Glucobay
- Group 2: Metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Bay G5421 Glucobay — Oral, dosage of Acarbose as per the directions of treating physician
  Groups: Group 1
Drug: Metformin — Oral, dosage of Metformin as per the directions of treating physician
  Groups: Group 2

SUMMARY:
The study is designed as non interventional to collect data on the effectiveness of acarbose and metformin monotherapy, respectively, in terms of change from baseline in post prandial blood glucose level at the end of 16 weeks in drug-naïve type 2 diabetic patients within each carbohydrates consumption subgroup under real-life treatment condition in large sample of type-2 diabetes patients in India. The study will begin after the study approval by ethics committee.All drug naïve patients in whom decision to administer acarbose or metformin monotherapy for type 2 diabetes management has been made will be included in study after taking the informed consent.Patients will be observed for up to 16 weeks (2 weeks).The study involves general examination of patients, collection of data like history of disease, concomitant medication, drug dose , 24 hr dietary recall etc. The study is planned to enroll 12250 subjects from multiple study centers spread across India. The study data will be analyzed with appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Drug-naïve (i.e., the patients should never be treated with anti-diabetic drugs before screening) patients in whom decision to administer monotherapy with either acarbose or metformin for type-2 diabetes management has been made by the attending physician on the basis of best clinical practice and medical patient needs, and who consent to participate in study will be included

Exclusion Criteria:

* Patients receiving any anti-diabetic medication at the time of enrollment in the study will be excluded. However, during observation period, patients may receive any additional anti-diabetics medication at the decision of investigator.
* Exclusion criteria should be read in conjunction with local product information. All contra-indications according to the local marketing authorization should be considered

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Drug-naïve sub-optimally controlled (by diet and physical exercise) type 2 diabetic patients (Female and male patients who are at least 18 years of age) selected from secondary or tertiary referral centers, private hospitals / clinic with good inflow of patients with diabetes
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The mean change in post-meal glucose levels from baseline at the end of observation period of up to 16 weeks | baseline and 16 weeks
  The primary outcome will be summarized separately in acarbose and metformin monotherapy treated patients having carbohydrates consumption (National Institute of Nutrition (NIN), India recommend50% to 60% of total calories from carbohydrates in balance diet : - Below NIN recommendation (< 50%) - As per NIN recommendation (50% to 60%) - Above NIN recommendation (> 60%)

SECONDARY OUTCOMES:
Mean change of HbA1c | Baseline and 16 weeks
Mean change of fasting blood glucose(FBG) | Base line and 16 weeks
Mean change of low density lipoprotein cholesterol(LDL) | baseline and 16 weeks
Mean change of high density lipoprotein cholesterol(HDL) | Baseline and 16 weeks
Mean change of total cholesterol(TC) | baseline and 16 weeks
Mean change of Body weight | baseline and 16 weeks
Mean change of triglyceride(TG) | baseline and 16 weeks
Compare the mean change between acarbose and metformin arm of postprandial blood glucose (PPBG) | baseline and 16 weeks
Compare the mean change between acarbose and metformin arm of HbA1c | baseline and 16 weeks
Compare the mean change between acarbose and metformin arm of FBG | baseline and 16 weeks
Compare the mean change between acarbose and metformin arm of LDL | baseline and 16 weeks
Compare the mean change between acarbose and metformin arm of HDL | baseline and 16 weeks
Compare the mean change between acarbose and metformin arm of TC | baseline and 16 weeks
Compare the mean change between acarbose and metformin arm of TG | baseline and 16 weeks
Compare the mean change between acarbose and metformin arm of Body weight | baseline and 16 weeks
Change in gastrointestinal tolerability to therapy from post baseline visit to the end of observation period of up to 16 weeks | baseline and 16 weeks
Incidence rate of adverse drug reactions in acarbose and metformin treated groups during 16 weeks observation period | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer